CLINICAL TRIAL: NCT04585490
Title: Personalized Escalation of Consolidation Treatment Following Chemoradiotherapy and Immunotherapy in Stage III NSCLC
Brief Title: Personalized Escalation of Consolidation Treatment Following Chemoradiotherapy and Immunotherapy in Stage III NSCLC in Stage III NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Maximilian Diehn (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Maximilian Diehn, Vice Chair of Research, Division Chief of Radiation and Cancer Biology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-54807; LUN0114 (Other: OnCore); NCI-2021-09500 (Other: Clinical Trial Reporting Program)
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer; NSCLC, Stage III; Nsclc
Keywords: durvalumab; tremelimumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Carboplatin; Pemetrexed; Glutamic Acid; Paclitaxel; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Cohort 1 minimal residual disease positive (MRD+) (Experimental): Subjects with detectable ctDNA will receive 4 cycles of platinum doublet chemotherapy [carboplatin/pemetrexed], tremelimumab (75 mg IV every 21 days) and durvalumab (1500 mg IV every 21 days), except subjects with squamous cell carcinoma histology will receive carboplatin/paclitaxel. Subjects will be evaluated with PET/CT and/or computed tomography (CT) thorax every 12 weeks. Following ctDNA evaluation, in the absence of progression or toxicity, subject will continue with durvalumab to complete 1 year of treatment as standard of care.
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Cisplatin; Device: AVENIO ctDNA Surveillance Kit; Drug: Tremelimumab
- Cohort 2 minimal residual disease negative (MRD ) (Experimental): Subjects with undetectable ctDNA at study enrollment will receive standard of care durvalumab (10 mg/kg every 2 weeks, or equivalent, for 1 year). If subjects in Cohort 2 MRD progress prior to close of study, blood will be drawn for ctDNA testing.
  Interventions: Drug: Durvalumab; Device: AVENIO ctDNA Surveillance Kit

INTERVENTIONS:
Drug: Durvalumab — Cohort 1 (1500 mg IV every 21 days, for 1 year), •Cohort 2 (10mg/kg every 2 weeks for 1 year)
  Other Names: Imfinzi; MEDI-4736; MEDI4736
Drug: Carboplatin — Target area under the curve (AUC) not to exceed 750mg on Day 1 of every 21-day cycle
  Other Names: Carboplat; Carbosol; Carboplatino; cis-diammine(cyclobutane-1,1-dicarboxylato)platinum
  Arms: Cohort 1 minimal residual disease positive (MRD+)
Drug: Pemetrexed — 500mg/m2 on Day 1 of every 21-day cycle
  Other Names: Alimta; MTA; LY231514; L-glutamic acid, N-(4-(2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo(2,3-d)pyrimidin-5-yl)ethyl)benzoyl)
  Arms: Cohort 1 minimal residual disease positive (MRD+)
Drug: Paclitaxel — 175mg/m2 on Day 1 of every 21-day cycle
  Other Names: Praxel
  Arms: Cohort 1 minimal residual disease positive (MRD+)
Drug: Cisplatin — Cisplatin (75mg/m2 per institution guidelines) may be substituted for Carboplatin
  Other Names: platinum diamminodichloride; Abiplatin; Cismaplat; cis-platinum; Platinex; platinum, diaminedichloro-, cis- (8CI)
  Arms: Cohort 1 minimal residual disease positive (MRD+)
Device: AVENIO ctDNA Surveillance Kit — Roche Sequencing and Life Science kit to detect minimal residue disease (MRD)
Drug: Tremelimumab — not to exceed 75mg IV on Day 1 of every 21-day cycle
  Other Names: Imjudo; Tremelimumab-actl; Ticilimumab; CP-675; CP-675,206
  Arms: Cohort 1 minimal residual disease positive (MRD+)

SUMMARY:
The purpose of this study is to test whether or not number of circulating cancer cells detected in the blood can be decreased the by combining the standard treatment (durvalumab) with Tremelimumab and additional chemotherapy

DETAILED DESCRIPTION:
Primary objective is to measure the change in the levels of circulating tumor DNA (ctDNA) in Cohort 1 (MRD+) due to the addition of Tremelimumab and platinum doublet chemotherapy in subjects with stage III unresectable disease with positive DNA treated with consolidation chemotherapy and immunotherapy.

Secondary Objectives:

To determine the proportion of subjects in Cohort 1 MRD+ for whom ctDNA becomes undetectable after adding chemotherapy and tremelimumab to consolidation durvalumab

To describe compare overall survival (OS) of subjects with baseline detectable ctDNA (Cohort 1 MRD+) vs baseline undetectable ctDNA (Cohort 2 MRD ) ·To compare progression free survival (PFS) between subjects with baseline detectable (Cohort 1 MRD+) vs baseline undetectable ctDNA (Cohort 2 MRD )

ELIGIBILITY:
Inclusion Criteria:

1. Histologically- or cytologically-documented NSCLC presenting with locally-advanced, unresectable stage III disease (Version 8 of AJCC Staging Manual) or NSCLC with locoregional recurrence after previous definitive treatment.
2. For stage III or recurrent disease, must have completed platinum-based chemotherapy and radiation therapy to all known tumor sites (60 Gy +/- 10%). Must not have known progression of disease.
3. Must be receiving consolidation durvalumab following completion of radiation and chemotherapy, and less than 32 weeks has elapsed from their first dose of durvalumab. (Patients may sign consent for study before start of durvalumab, but confirm eligibility and enroll only after first dose of durvalumab is received).
4. Able to potentially receive further consolidation chemotherapy plus durvalumab and tremelimumab, but not be currently intended to receive additional systemic consolidation chemotherapy apart from this durvalumab.
5. Pre-treatment tumor tissue or tumor DNA sample is believed to be available for analysis
6. Aged 18 years or older
7. Weight > 30kg
8. Life expectancy ≥ 12 weeks
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
10. Absolute neutrophil count > 1.0 x 109/L (1000/mm3)
11. Platelets > 75 x 109/L (100,000/mm3)
12. Hemoglobin ≥ 9.0 g/dL (5.59 mmol/L)
13. Measured creatinine clearance > 40 mL/min, by either 24 hour urine collection or the Cockcroft Gault formula

    Males:

    Mass(kg) x (140-Age) / 72 x serum creatinine (mg/dL)

    Females:

    Mass(kg) x (140-Age) x 0.85 / 72 x serum creatinine (mg/dL)
14. Serum bilirubin ≤ 1.5 x upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of evidence of hemolysis or hepatic pathology) who will be allowed in consultation with their physician.
15. aspartate aminotransferase (AST) (SGOT)/Alanine Aminotransferase (ALT) (SGPT) ≤ 2.5 x institutional upper limit of normal (ULN) unless liver metastases are present, in which case it must be ≤ 5 x ULN
16. Ability to understand and the willingness to sign the written IRB approved informed consent document.

Exclusion Criteria:

Involvement in the planning and/or conduct of the study

2. Previous enrollment or randomization in the present study

3. Received Investigational product as part of another clinical study

4. Mixed small cell and non small cell lung cancer histology

5. History of another primary malignancy and currently undergoing active treatment.

Exception: May participate if receiving adjuvant endocrine therapy for breast or prostate cancer.

6. Current or prior use of immunosuppressive medication within 14 days before enrollment, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for locally advanced NSCLC is allowed.

7. Any unresolved toxicity CTCAE > Grade 2 from the prior chemoradiation therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

* Subjects with Grade ≥ 2 neuropathy will be evaluated on a case by case basis after consultation with the Protocol Director / Principal Investigator
* Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by treatment with durvalumab may be included (ie, hearing loss) only after consultation with the Protocol Director / Principal Investigator.

  8. Any prior Grade ≥ 3 immune related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > Grade 1) that may limit subject from continuing durvalumab during the study

  9. Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) that would prevent administration of study drug.

  10. Active or prior documented autoimmune or inflammatory disorders which is likely to limit the subjects ability to continue durvalumab on the study (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis; Graves' disease; rheumatoid arthritis; hypophysitis; uveitis; etc]). Those with history of autoimmune or inflammatory disorders who are currently tolerating durvalumab may be eligible to participate with approval from the PI. The following are also exceptions to this criterion:
  1. Vitiligo or alopecia
  2. Hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
  3. Chronic skin condition not requiring systemic therapy
  4. Celiac disease controlled by diet alone

     11. History of primary immunodeficiency

     12. History of organ transplant requiring therapeutic immunosuppression

     13. History of hypersensitivity to carboplatin, pemetrexed, paclitaxel, or nab-paclitaxel that is likely to prevent re-administration of these agents

     14. Active infection including but not limited to:
* Grade 3 or higher clinically significant infection
* Active known Hepatitis B [known positive results for HBV surface antigen (HBsAg) within 2 months prior to enrollment]. EXCEPTION: Subjects with a past or resolved HBV infection, defined as the presence of hepatitis B core antibody (anti-HBc) and absence of HBsAg are eligible
* Active known Hepatitis C (HCV). EXCEPTION: Subjects positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA
* Active known tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
* Active known HIV infection

  15. Receipt of live attenuated vaccine within 30 days prior to the first dose of concurrent chemotherapy and durvalumab. Note: Subjects, if enrolled, should not receive live vaccine through 30 days after the last dose of chemotherapy concurrent with durvalumab.

  16. Uncontrolled intercurrent illness, including but not limited to:
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Uncontrolled hypertension
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Interstitial lung disease
  * Serious chronic gastrointestinal conditions associated with diarrhea
  * Psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent.

    17. Female subjects who are pregnant or breast feeding; or subjects of reproductive potential of any gender who are not employing or who do not agree to employ an effective method of birth control prior to trial enrollment.ollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in ctDNA Level Following Chemotherapy | 12 weeks
  Participants in Cohort 1 MRD+ will be assessed for ctDNA levels at baseline and end of treatment, expected to be 4 cycles of 3 weeks per cycle (defined as ctDNA evaluable set or ctDES). The outcome will be assessed as the number of participants with a ≥ 3 fold decrease in ctDNA level, a number without dispersion.

SECONDARY OUTCOMES:
Presence of Detectable ctDNA Following Chemotherapy | 12 weeks
  Participants in Cohort 1 MRD+ will be assessed for ctDNA levels at baseline and end of treatment, expected to be 4 cycles of 3 weeks per cycle. The outcome will be assessed as the number of participants with or without detectable ctDNA, a number without dispersion.
Overall Survival (OS) | 2 years
  Overall survival (OS) is defined as the period a participant remains alive after study registration until death due to any cause. Participants lost to follow up will be censored at last known date alive. The outcome will be reported as the number of participants in both cohorts remaining alive after 2 years, a number without dispersion.
Progression free survival (PFS) | 2 years
  Progression free survival (PFS) is defined as the period a participant remains alive without disease progression after study registration. Tumor status is assessed per the Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) by computed tomography (CT), positron emission tomography (PET) CT; and/or X rays. Participants lost to follow up will be censored at last known date alive. The outcome will be reported as the number of participants in both cohorts remaining alive without progression after 2 years, a number without dispersion.
  * Complete Response (CR) = Disappearance of all lesions
  * Partial Response (PR) = ≥30% decrease in the sum of the lesion diameters
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of lesion diameters, and/or the appearance of 1+ new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Durvalumab and Tremelimumab related Adverse Events (Cohort 1 MRD+ only) | 13 months
  Adverse events will be collected for participants of Cohort 1 (MRD+) who initiate treatment with durvalumab and tremelimumab through 930 days after the last dose of durvalumab. AE grade per the Common Terminology Criteria for Adverse Events (CTCAE v5) criteria and relationship to study treatment will be assessed. The outcome will be reported as the number of durvalumab and tremelimumab related adverse events by grade that Cohort 1 MRD+ participants experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Diehn, MD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No